CLINICAL TRIAL: NCT00735579
Title: Incidence of Wound-healing-abnormalities in Major Abdominal Surgery - Association With Factors of Coagulation
Brief Title: Wound Healing Abnormalities in Major Abdominal Surgery
Acronym: INWOUND
Status: Completed | Type: Observational
Sponsor: Klinikum St. Georg gGmbH (Other)
Responsible Party: Principal Investigator, Armin Sablotzki, MD, Prof. Dr. med., Klinikum St. Georg gGmbH
Other Study IDs: EK-BR-21/08-1; Stu08/0022
Record Dates: First submitted 2008-08-14; First posted 2008-08-15 (Estimated); Last update posted 2017-04-24 (Actual); Status verified 2017-04

CONDITIONS: Impaired Wound Healing; Factor XIII Deficiency
Keywords: major abdominal surgery; coagulation; extracellular matrix proteins; wound healing after major abdominal surgery
MeSH Terms: conditions — Factor XIII Deficiency; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 1) serum samples for measurement of coagulation factors
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study group: Patients undergoing major abdominal surgery

SUMMARY:
This clinical observational study investigates the incidence of wound healing abnormalities in patients undergoing major abdominal surgery. Second aim of the study is, if wound healing deficits may be accompanied by abnormalities in blood coagulation parameters.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Male or female
* Informed consent
* Major abdominal surgery

Exclusion Criteria:

* Pre-existing coagulation abnormalities
* Pre-existing severe renal or liver failure
* Chemo- or radiochemotherapy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing major abdominal surgery
Sampling Method: Non-Probability Sample
Enrollment: 260 (Actual)
Dates: Start 2008-07; Primary Completion 2017-04-21 (Actual); Study Completion 2017-04-21 (Actual)

PRIMARY OUTCOMES:
Incidence of wound healing abnormalities | from baseline to postoperative day 28
  Occurence of wound healing abnormalities within the first 28 days after surgery

SECONDARY OUTCOMES:
Abnormalities in coagulation parameters | postoperative day 28
  occurence of low platelets (<60.000) or factor XIII < 50% between the first and seventh postoperative day

CONTACTS AND LOCATIONS:
Overall Officials: Armin R Sablotzki, MD, Principal Investigator — Klinikum St. Georg gGmbH
Locations (1):
- Klinikum St. Georg gGmbH, Leipzig, Saxony, Germany

REFERENCES:
- See also: Related Info — http://www.sanktgeorg.de